CLINICAL TRIAL: NCT05862051
Title: Randomised Phase II Trial to Evaluate Progression-Free Survival in Integrating Local Ablative Therapy With First-Line Systemic Treatment for Unresectable Oligometastatic Colorectal Cancer
Brief Title: RESOLUTE Trial Aims to Investigate the Value of Adding Local Ablative Treatment to Standard Systemic Treatment for Unresectable Oligometastatic Colorectal Cancer
Acronym: RESOLUTE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Australasian Gastro-Intestinal Trials Group (Network)
Collaborators: Walter and Eliza Hall Institute of Medical Research (Other); Cancer Council Victoria (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RESOLUTE
Record Dates: First submitted 2022-12-08; First posted 2023-05-17 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Colorectal Cancer; Oligometastatic Disease
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Local ablative therapies (LAT) arm (Experimental): A maximum of three Local ablative therapy (LAT) modalities can be administered for each participant, with a maximum of 2 modalities per organ, provided all LAT can be delivered within 12 weeks and participant can safely resume systemic treatment within 16 weeks from randomisation.
  After completing LAT, participant is to resume a further two to three months of first-line systemic treatment to a total of 6 months (including the initial 3-4 months of treatment). For patients receiving a doublet or triplet regimen, treatment may be de-escalated to maintenance fluoropyrimidine +/- biologics or anti-EGFR monotherapy at any point after trial entry at clinician discretion. The treating clinician may choose to discontinue systemic treatment following LAT for patients who have experienced prior intolerable toxicity.
  Interventions: Procedure: Local Ablative Therapy; Procedure: Standard first-line systemic treatment
- Control arm (Placebo Comparator): The first-line systemic treatment will be standard of care as determined by the treating clinician. The following standard chemotherapy regimens are allowed: single agent fluoropyrimidine, CAPOX, FOLFOX, FOLFIRI, CAPIRI or FOLFOXIRI. Treatment with a biologic is allowed including bevacizumab or an anti-EGFR antibody (cetuximab or panitumumab). For patients receiving a doublet or triplet regimen, treatment may be de-escalated to maintenance fluoropyrimidine +/- biologics or anti-EGFR monotherapy at any point after trial entry at clinician discretion.
  Interventions: Procedure: Standard first-line systemic treatment

INTERVENTIONS:
Procedure: Local Ablative Therapy — LAT modalities allowed include surgical resection, stereotactic radiotherapy (SRT), laparoscopic or percutaneous thermal ablation [radiofrequency ablation (RFA) or microwave ablation (MWA)]. The LAT modalities will be delivered by specialists in the field (surgeons, radiation oncologists and/or interventional radiologists). The precise mode of delivery and number of times the LAT modality is delivered is case-dependent and is determined at a multi-disciplinary meeting (MDM).
  Arms: Local ablative therapies (LAT) arm
Procedure: Standard first-line systemic treatment — Standard of care as determined by the treating clinician. The following standard chemotherapy regimens are allowed: single agent fluoropyrimidine, CAPOX, FOLFOX, FOLFIRI, CAPIRI or FOLFOXIRI. Treatment with a biologic is allowed including bevacizumab or an anti-EGFR antibody (cetuximab or panitumumab). For patients receiving a doublet or triplet regimen, treatment may be de-escalated to maintenance fluoropyrimidine +/- biologics or anti-EGFR monotherapy at any point after trial entry at clinician discretion.

SUMMARY:
This study aims to assess the clinical benefit of local ablative therapy (LAT) following initial standard first-line systemic treatment including the impact on survival, compared to continued standard first-line systemic treatment for oligometastatic colorectal cancer.

DETAILED DESCRIPTION:
Who is this study for:

Adults with unresectable oligo-metastatic colorectal who have demonstrated treatment benefit (partial response or stable disease as per RECIST criteria) after 3-4 months of standard first-line systemic treatment.

Study details

Participants will be randomly allocated to either a LAT arm, who will receive metastasis-directed LAT such as radiotherapy or thermal ablation following initial standard first-line systemic treatment, or a control arm who will receive continued first-line systemic treatment alone. Those receiving LAT will return to systemic treatment 16 weeks post-randomisation. Information on progression-free survival and treatment outcomes will be collected.

Data from this study will inform investigators of the potential benefit of local ablative therapy in the therapeutic setting for metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic colorectal adenocarcinoma that is not amenable to potentially oncological curative surgery alone.
* Primary tumour must be controlled if the primary is intact, with no evidence of progression at primary site prior to study entry
* Imaging demonstrating ongoing treatment benefit (partial response or stable disease as per RECIST criteria) after 3-4 months of standard first-line systemic treatment.
* At least one metastatic lesion detected on CT +/- FDG-PET scan prior to first line systemic treatment AND on screening FDG-PET and CT scans, meeting the following criteria:

  1. max of 3 lesions per organ except for the liver and lung
  2. max of 5 lesions in the lung
  3. no limitation to the number of liver lesions provided they are all amenable to LAT
  4. max of 3 involved organs including a lymph node station
  5. only one lymph node station involvement is allowed
  6. for patients with liver metastases, a quadruple phase contrast enhanced CT or MRI liver is required to fully stage the liver; this can be performed prior to or within 4 weeks of commencing first line systemic treatment
  7. staging FDG-PET scan is encouraged and can be performed prior to or within 4 weeks of commencing first line systemic treatment
* All lesions can be safely treated by LAT as determined by multidisciplinary team meeting.

Exclusion Criteria:

* Deficient mismatch repair (dMMR) or microsatellite instability-high (MSI-high) tumour
* BRAFV600E mutated tumour
* Concurrent or previous other malignancy within 2 years of study entry, except curatively treated basal or squamous cell skin cancer, prostate intraepithelial neoplasm, carcinoma in-situ of the cervix, Bowen's disease or prostate cancer with a Gleason score ≤6.
* Presence of brain, peritoneal, omental or ovarian metastases
* Malignant pleural effusion or ascites.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2021-12-14 (Actual); Primary Completion 2024-06-14 (Estimated); Study Completion 2025-06-14 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 12 Months from randomisation
  To compare the efficacy of metastasis-directed LAT following initial standard first-line systemic treatment vs continued first-line systemic treatment alone, as measured by Progression-Free Survival (PFS)

SECONDARY OUTCOMES:
Overall survival | 12 Months from randomisation and through study completion, an average of 1 year
  To compare the efficacy of LAT following initial standard first-line systemic treatment, compared to continued first-line systemic treatment alone, as measured by Overall Survival (OS)
Efficacy of local ablative therapy | 12 Months from randomisation and through study completion, an average of 1 year
  To compare the efficacy of LAT following initial standard first-line systemic treatment, compared to continued first-line systemic treatment alone, on:
  1. time to development of new metastatic lesions.
  2. time to initiation of 2nd line systemic treatment.
Time to progression following local ablative therapy | Through study completion, an average of 1 year
  To assess the time to progression of LAT treated lesions.
Systemic treatment-free interval | Through study completion, an average of 1 year
  To compare systemic treatment-free interval between the two treatment groups.
Rate of high-grade toxicities | Through study completion, an average of 1 year
  To assess and compare rate of high-grade (Grade 3-5) toxicities between the two treatment groups.
Quality of life measure | Through study completion, an average of 1 year
  To compare quality of life measures between the two treatment groups using patient questionnaire - The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) using the 4-point ordinal scale (not at all, a little, quite a bit and very much)

CONTACTS AND LOCATIONS:
Locations (9):
- Australia (9):
  - Border Medical Oncology, Albury, New South Wales
  - Bendigo Hospital, Bendigo, Victoria
  - Eastern Health, Box Hill, Victoria
  - The Northern Hospital, Epping, Victoria
  - St Vincent's Hospital Melbourne, Fitzroy, Victoria
  - Peter MaCallum Cancer Centre, Melbourne, Victoria
  - Peninsula Health, Rosebud, Victoria
  - Western Health, Saint Albans, Victoria
  - Northeast Health Wangaratta, Wangaratta, Victoria

IPD SHARING:
Plan to Share IPD: No